CLINICAL TRIAL: NCT01794871
Title: The Histological Analysis in Renal Transplantation Patients With Deterioration of Graft Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COLO400ACN03T
Record Dates: First submitted 2013-02-16; First posted 2013-02-20 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Allograft Dysfunction

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — graft biopsy after kidney transplantation
Oversight: Data Monitoring Committee: No

SUMMARY:
Identify the cause of chronic allograft dysfunction using a combination of comprehensive clinical and histologic information in Chinese renal transplant recipients, then to identify the position of CNI nephrotoxicity in CAD.Chronic allograft dysfunction reflects the dual impact of both immunologic and nonimmunologic (primarily calcineurin inhibitor [CNI]nephrotoxicity) injury. In previous, CNI nephrotoxicity is overstated and considered one of the major causes of CAD, however, recently there has been found most death-censored graft losses to be the result of alloimmune or autoimmune injury, with only a minority of cases attributable to CNI toxicity. Unfortunately, Situation of objective CNI toxicity in CAD in China is not well analyzed. To improve perception of Neo safety with more local evidence, we want to do a retrospective study to identify the cause of chronic allograft dysfunction using a combination of comprehensive clinical and histologic information in Chinese renal transplantation recipients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Kidney transplant recipients, only including recipients of living-donor grafts
* Underwent an allograft biopsy between January 2005 and December 2011 because of developing deterioration of graft function*.

  * Deterioration of function was defined as (1) an unexplained and persistent greater than or equal to 25% increase of CR over baseline (in the absence of potential confounding factors) or (2) new onset proteinuria (defined as albumin/CR ratio ≥0.2 or a protein/CR ratio >0.5).

Exclusion Criteria:

* Multiple organ transplants, prior transplant with any other organ or tissue
* Patients who did not have the information regarding the pathological diagnosis
* Patients who did not have the histological sections of the allograft biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Maintenance living donor renal transplant recipients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-03 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
the graft biopsy of maintenance living donor renal transplant recipients who underwent deterioration of graft function | up to 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China